CLINICAL TRIAL: NCT05324332
Title: A Pilot Comparison of 68Ga-P16-093 and 68Ga-PSMA-11 in the Same Group of Primary Prostate Cancer Patients
Brief Title: 68Ga-P16-093 and 68Ga-PSMA-11 PET/CT Imaging in the Same Group of Primary Prostate Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH P16-093
Record Dates: First submitted 2022-04-03; First posted 2022-04-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-P16-093 and 68Ga-PSMA-11 PET/ CT scan (Experimental): Patients of Prostate cancer PET/CT imaging: In two consecutive days, each patient underwent whole-body PET/CT scan after intravenous administration of 68Ga-P16-093 and 68Ga-PSMA-11, respectively.
  Interventions: Drug: 68Ga-P16-093; Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 68Ga-P16-093 — Intravenous injection of 68Ga-P16-093 with the dosage of 1.8-2.2 MBq (0.05-0.06 mCi)/kg. Tracer doses of 68Ga-P16-093 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: 68Ga-P16-093 injection
Drug: 68Ga-PSMA-11 — Intravenous injection of 68Ga-PSMA-11 with the dosage of 1.8-2.2 MBq (0.05-0.06 mCi)/kg. Tracer doses of 68Ga-PSMA-11 will be used to image lesions of prostate cancer by PET/CT.
  Other Names: 68Ga-PSMA-11 injection

SUMMARY:
Prostate-specific membrane antigen (PSMA)-targeted PET imaging with 68Ga-labeled compounds is able to provide superior sensitivity and specificity to detect primary prostate tumor and its metastases, like the most widely studied 68Ga-PSMA-11. This pilot study was evaluate the diagnostic performance of 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, which was compared with 68Ga-PSMA-11 in the same group of primary prostate cancer patients.

DETAILED DESCRIPTION:
Prostate cancer (PC) is one of the most common malignancies worldwide in men, with persistently high numbers dying from this disease. Due to low levels of glycolysis in prostate cancer cell, the uses of 18F-FDG PET/CT to detect prostate cancer and its metastases are limited. Prostate specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. Various low molecular weight radiopharmaceuticals targeting PSMA such as PSMA-11, PSMA-617 for 68Ga-labeling have been developed. 68Ga-PSMA PET/CT has demonstrated desirable sensitivity and specificity in the detection of prostate cancer lesions, which can find many micro lesions that cannot be identified by CT, MRI and bone scan. 68Ga-P16-093, a novel radiopharmaceutical modified based on 68Ga-PSMA-11, with the urea fragment of a conjugate that employs the HBED-CC chelator for labeling with 68Ga(III). The HBED-based chelating ligand binds the 68Ga3+ ion with high affinity in a pseudo-octahedral N2O4 coordination sphere by its two phenolate O, two amino-acetate carboxylate O, and two amino N donor atoms. This pilot study was prospectively designed to evaluate the diagnostic performance of 68Ga-P16-093 compared with 68Ga-PSMA-11 in the same group of primary prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed untreated primary prostate cancer patients;
* 68Ga-PSMA-11 and 68Ga-P16-093 PET/CT within a week;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor detection rate | through study completion, an average of 1 year
  comparing the number of tumor detected by 68Ga-P16-093 and 68Ga-PSMA-11 PET/CT

SECONDARY OUTCOMES:
standardized uptake value (SUV) of tumor | through study completion, an average of 1 year
  comparing the SUVmax of tumor derived from 68Ga-P16-093 and 68Ga-PSMA-11 PET/CT

OTHER OUTCOMES:
PSMA expression and SUV | through study completion, an average of 1 year
  Correlation between PSMA immunoreactive score and SUVmax of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang J, Li L, Chen J, Wang R, Xiang J, Peng X, Wang Y, Luo Y, Zhu L, Kung HF, Zhou Z, Xiao Y, Zhu Z. [68Ga]Ga-P16-093 PET/CT in newly diagnosed prostate cancer: Histopathological validation and comparison with [68Ga]Ga-PSMA-11. Eur J Nucl Med Mol Imaging. 2025 Dec 10. doi: 10.1007/s00259-025-07687-0. Online ahead of print. PMID 41366119
- [Derived] Wang G, Li L, Zhu M, Zang J, Wang J, Wang R, Yan W, Zhu L, Kung HF, Zhu Z. A prospective head-to-head comparison of [68Ga]Ga-P16-093 and [68Ga]Ga-PSMA-11 PET/CT in patients with primary prostate cancer. Eur J Nucl Med Mol Imaging. 2023 Aug;50(10):3126-3136. doi: 10.1007/s00259-023-06283-4. Epub 2023 May 26. PMID 37233785